CLINICAL TRIAL: NCT04229810
Title: Individualized Perioperative Open Lung Ventilatory Approach in Emergency Abdominal Laparotomy. A Prospective Multicenter Randomized Controlled Trial.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Carlos Ferrando Ortolá, Head of Surgical Intensive Care Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: iPROVE-EAL
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Ventilator Lung

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STD-02 (Active Comparator): Conventional standardized lung protective ventilation.
  Interventions: Procedure: STD-02
- iOLA-iHFNC (Experimental): Individualized ventilatory strategy that mantains an open lung condition.
  Interventions: Procedure: iOLA-iHFNC

INTERVENTIONS:
Procedure: STD-02 — Conventional standardized ventilatory approach.
  Arms: STD-02
Procedure: iOLA-iHFNC — Indivudualized perioperative open lung ventilatory approach.
  Arms: iOLA-iHFNC

SUMMARY:
Prospective multicenter randomized controlled trial. Individualized perioperative open lung ventilatory approach in emergency abdominal laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women ≥18 years of age who underwent emergency laparotomy with the presence of post-induction positive air-test (SpO2 <97% after a maximum of 15 minutes at FIO2 of 0.21). A SpO2 <97% at any FIO2 would also be considered a positive air-test.

Exclusion Criteria:

* 1) Pregnancy or breast feeding, 2) Moderate or severe ARDS defined, 3) refractory shock, 4) diagnosis or suspected intracranial hypertension (>15mmHg), 5) mechanical ventilation in the last 15 days (including CPAP), 6) presence of pneumothorax or giant bullae in a chest radiograph or computed tomography (CT), 7) patients participating in another intervention study with the same or similar primary outcome variable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Severe postoperative pulmonary complications | 7 days
  A composite of severe postoperative pulmonary complications appearing during the first 7 postoperative days. Postoperative pulmonary complication will include any of the following: 1) Respiratory failure, 2) Pneumothorax, 3) Weaning failure, 4) Acute respiratory distress syndrome (ARDS), 5) Pulmonary infection.

IPD SHARING:
Plan to Share IPD: No